CLINICAL TRIAL: NCT05371587
Title: The Effects of the Autonomy and Perceptions Approach to Resistance Training (APART) on Body Composition, Physiological and Performance Outcomes in Healthy Young Adults: a Non-inferiority Randomized Controlled Trial
Brief Title: The Effects of Autonomy and Perceptions on Resistance Training Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Israel Halperin, Principle investigator, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISF_Halperin_TAU
Record Dates: First submitted 2022-05-01; First posted 2022-05-12 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-08

CONDITIONS: Strength Training
Keywords: Autonomy; Perception of effort

STUDY DESIGN:
Intervention Model Description: A parallel two-armed, non-inferiority randomized controlled trial
Who Masked: Participant
Masking Description: Participants are allocated using sealed envelops, they receive their arm identification "A" or "B" without information regarding the intervention or group differences. Data will be analyzed using the identification letter without treatment allocation information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A - Standard resistance training prescription (Active Comparator): Standard resistance training prescription: participants will perform three sessions per week comprised of six resistance training exercises - horizontal leg press, lat-pulldown, knee extension, chest press, leg curls and shoulder press. They will perform 3 sets of 10 repetitions using 65% percent of the maximal load that can be lifted once according to a one repetition maximum (1RM) test. Their progression model will be as follows:
  Weeks 1-3 65%1RM; Weeks 4-6 70%1RM; 1RM reassessment at week 6; Weeks 7-9 70% of the updated 1RM; Weeks 10-12 75%1RM.
  Prior to beginning of the program four visits will take place:
  1. Laboratory visit for measuring physiological and anthropometric outcomes (see outcomes section)
  2. 1RM testing
  3. Endurance and maximal voluntary contraction testing + introduction with the exercise program
  4. A second introduction session with the exercise program
  Interventions: Other: Standard prescription
- B- Autonomy and perceptions approach to resistance training (APART) (Experimental): Participants will perform 3 sessions/week of the same exercises. They will perform 3 sets of each exercise, self-select the load they lift in each set and perform repetitions aiming to reach a level of effort of 7-8 on a 0-10 rating of perceived effort scale (RPE) at the end of the set. Their progression model will be as follows: Weeks 1-3 RPE 7/10; Weeks 4-12 RPE 8/10. The selected RPE score of 7 and then 8 out of 10 has been shown to lead to increases in maximal strength in previous research. Prior to beginning of the program four visits will take place:
  1. Laboratory visit (similar to standard).
  2. 1RM testing where the principles of perceived effort will be introduced.
  3. Endurance and maximal voluntary contraction testing + introduction with the exercise program. Participants will practice how to self-select the load they prefer and then perform repetitions leading to the target RPE score.
  4. A second introduction session with the exercise program and the RPE construct.
  Interventions: Other: Autonomy and Perceptions Approach to Resistance Training (APART)

INTERVENTIONS:
Other: Autonomy and Perceptions Approach to Resistance Training (APART) — Alternative resistance training prescription based on trainees' autonomy and perceptions.
  Arms: B- Autonomy and perceptions approach to resistance training (APART)
Other: Standard prescription — Standard resistance training prescription, based on international organization's guidelines.
  Arms: A - Standard resistance training prescription

SUMMARY:
120 participants will be randomized into one of two groups that will perform resistance training at a gym three time per week for three months. One group will follow common resistance training guidelines, whereas the other will exercise according to their preferences and perception of effort. The groups will be compared on the following primary outcomes after six and 12 weeks: body composition, physiological and performance tests. The groups will be compared on the following secondary outcomes every two weeks: enjoyment and satisfaction levels. Adherence rates will be measured throughout the intervention.

DETAILED DESCRIPTION:
Develop and test the non-inferiority of a new RT prescription model, entitled The Autonomy and Perceptions Approach to Resistance Training (APART). This approach is simple to follow, individualized, and autonomy supportive. Accordingly, it may assist trainees to overcome some of the limitations of the standard RT prescription approach. Under APART, trainees choose the loads they lift for each exercise according to their preferences, and then complete as many repetitions as required until reaching a specific rating of perceived effort (RPE) value on a 0 (no effort) to 10 (maximal effort) scale (e.g., 8/10). For this non-inferiority randomized controlled trial, the investigators will recruit 120 healthy, sedentary participants, between the ages of 18 and 45, who will be block-randomized by gender and age (18-27, 28-45) to either the APART or the standard groups. Following two baseline-testing sessions and two guided familiarization sessions, participants will independently complete three RT sessions per week for 12 weeks. The following primary outcomes will be assessed after six and 12 weeks: (ⅰ) body composition including fat free mass; (ⅱ) performance measures, including maximal strength and strength endurance; and (ⅲ) physiological measures, including blood profile and hemodynamics. The following secondary outcomes will be measured every two weeks: (ⅳ) psychological measures, including self-efficacy, autonomy, and enjoyment; and (ⅴ) adherence measures, which will be monitored throughout the intervention. If APART will be found to be non-inferior to the standard RT prescription, it can provide a simple and easy to follow alternative to the standard RT prescriptions, which also highlights trainees' preferences and individual abilities. This, in turn, might contribute to future participation and adherence to RT.

ELIGIBILITY:
Inclusion Criteria:

* No health issues preventing resistance training
* Body mass index (BMI) between 18.5 ("normal") and 29.9 ("overweight")
* Body weight > 50 Kg
* Without RT experience or with little experience (i.e. less than once a week in the past 12 months).

Exclusion Criteria:

* Participants who responded positively to any of the health sections and did not provide medical clearance
* Pregnant women or less than six months after childbirth
* BMI values outside of the specified range
* Body weight < 50 Kg
* RT experience exceeding the specified cut-off (see above)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure | Baseline to twelve weeks
  Participants will rest in a relaxed seating position for five minutes. Then their blood pressure and resting heart rate will be taken using an Omron M7 (HEM-780-E) blood pressure measuring device.
Change in Low Density Lipoprotein (LDL) value | Baseline to twelve weeks
  The blood samples will be collected by single-use disposable needle. A total of 20 mL of blood will be collected at each time-point in two, 10 mL Vacutainer® tubes: a plasma tube containing anticoagulant and a serum tube where the blood is allowed to clot. Plasma samples will be stored in ice until centrifuged twice at 1,500g for 10 minutes at 4° Celsius. Serum will be kept in room temperature for 60 minutes then centrifuged at 1300g for 10 minutes. Both samples will be divided into separate 1.8-mL microcentrifuge tubes and will be frozen at -80° C for later analysis.
Change in fasting glucose value | Baseline to twelve weeks
  The blood samples will be collected by single-use disposable needle. A total of 20 mL of blood will be collected at each time-point in two, 10 mL Vacutainer® tubes: a plasma tube containing anticoagulant and a serum tube where the blood is allowed to clot. Plasma samples will be stored in ice until centrifuged twice at 1,500g for 10 minutes at 4° Celsius. Serum will be kept in room temperature for 60 minutes then centrifuged at 1300g for 10 minutes. Both samples will be divided into separate 1.8-mL microcentrifuge tubes and will be frozen at -80° C for later analysis
Change in fat free mass | Baseline to twelve weeks
  Fat free mass will be measured using the SECA mBCA 515 (Seca, Hamburg, Germany), a valid and reliable analyzer of body composition. Participants will drink 400 ml of water before the examination which will take place in the morning. Drinking will be stopped 30 minutes before the examination and participants will be instructed to urinate and remove any jewelries before the examination.
Change in waist circumference | Baseline to twelve weeks
  Waist circumference will be measured according to WHO protocol: Participants will expose the area between their ribs and pelvic. The same investigator will measure the distance between the lower end of their ribcage and the anterior superior iliac spine (ASIS) and measure the waist circumference three times, midway between the two anatomical landmarks. The average value of the three measurements in centimeters will be documented for analysis.
Change in maximal muscle strength- One repetition maximum | Baseline to twelve weeks
  Participants will perform a dynamic warmup including mobility and calisthenics exercises, followed by specific warm up sets of each of the exercises: Horizontal leg press, knee extension and seated chest press (performed on weight-stack machines). Then, up to five attempts will be made to complete one repetition sets with increasing load until the participant either fails to complete the full range of motion or declares she cannot attempt the next set. The load (in kg) of the final successful attempt for each exercise will be documented for analysis. Two to three minutes rest will be provided between the attempts. The order of the exercises will be maintained throughout the assessment points and between participants. The assessments will be carried out by the same experimenter at the same time of day ±2 hours.
Change in muscle endurance | Baseline to twelve weeks
  Participants will perform a dynamic warmup including mobility and calisthenics exercises, followed by specific warm up sets of the knee extension and the chest press exercises. Then, 70% of the participant's identified maximal load (1RM) will be used to perform repetitions until task-failure (i.e., not able to complete another repetition). The number of completed repetitions will be documented for analysis. The same reference load will be used at six weeks. The order of the exercises will be maintained throughout the assessment points and between participants. The assessments will be carried out by the same experimenter at the same time of day ±2 hours.
Change in maximum voluntary contraction (MVC) - knee extension | Baseline to twelve weeks
  Isometric knee extension (using the knee extension machine) - will be assessed in a 90° angle using a link device (Kinvent, Link pull dynamometer) attached to a ratchet belt.

SECONDARY OUTCOMES:
Change in self efficacy questionnaire score | Baseline to twelve weeks
  The self-efficacy questionnaire is an eight items questionnaire. Respondents are required to read the statements and rate their level of agreement with each statement on a three points Likert scale. Score-range is 8-24. Higher scores indicate higher levels of self-efficacy.
Enjoyment | Six weeks to twelve weeks
  Participants will respond to an online survey examining their levels of enjoyment from the training sessions via a bi-polar scale ranging from -50 ("did not enjoy at all") to 50 ("extremely enjoyed").
Adherence | End of week 12
  Number of entries to the gym, documented by the gym front desk
Adherence without incentive | From week 12 to week 24
  Number of entries to the gym, documented by the gym front desk
Change in total cholesterol value | Baseline to twelve weeks
  The blood samples will be collected by single-use disposable needle. A total of 20 mL of blood will be collected at each time-point in two, 10 mL Vacutainer® tubes: a plasma tube containing anticoagulant and a serum tube where the blood is allowed to clot. Plasma samples will be stored in ice until centrifuged twice at 1,500g for 10 minutes at 4° Celsius. Serum will be kept in room temperature for 60 minutes then centrifuged at 1300g for 10 minutes. Both samples will be divided into separate 1.8-mL microcentrifuge tubes and will be frozen at -80° C for later analysis
Change in maximum voluntary contraction (MVC) - horizontal row | Baseline to twelve weeks
  Horizontal row (using the T-bar machine) - will be assessed in a 60° elbow angle using a link device (Kinvent, Link pull dynamometer) attached to a ratchet belt. Participants will lean their chest against the padded cushion with their feet stable on a designated built-in platform. They will pull the T-bar arm using a narrow grip. Their elbow angle will be measured using a goniometer. Then, three attempts will be made using 40%, 70% and 90% of their estimated MVC, followed by three attempts of 100% (i.e., MVC). 60 seconds rest will be provided between attempts. The average of the two high results will be documented for analysis.
Change in Hemoglobin | Baseline to twelve weeks
  The blood samples will be collected by single-use disposable needle. A total of 20 mL of blood will be collected at each time-point in two, 10 mL Vacutainer® tubes: a plasma tube containing anticoagulant and a serum tube where the blood is allowed to clot. Plasma tubes will be stored in ice and a complete blood count will be done within 60 minutes via Yumizen H500 analyzer.
Change in maximum voluntary contraction (MVC) - horizontal row | Baseline to twelve weeks
  Isometric horizontal row will be assessed in a 60° elbow flexion angle on the T-bar machine (Nautilus, WA, USA). The same link device will be secured using ratchet belts to match the desired setup for each participant.
Change in High Density Lipoprotein (HDL) value | Baseline to twelve weeks
  The blood samples will be collected by single-use disposable needle. A total of 20 mL of blood will be collected at each time-point in two, 10 mL Vacutainer® tubes: a plasma tube containing anticoagulant and a serum tube where the blood is allowed to clot. Plasma samples will be stored in ice until centrifuged twice at 1,500g for 10 minutes at 4° Celsius. Serum will be kept in room temperature for 60 minutes then centrifuged at 1300g for 10 minutes. Both samples will be divided into separate 1.8-mL microcentrifuge tubes and will be frozen at -80° C for later analysis.
Change in triglycerides value | Baseline to twelve weeks
  The blood samples will be collected by single-use disposable needle. A total of 20 mL of blood will be collected at each time-point in two, 10 mL Vacutainer® tubes: a plasma tube containing anticoagulant and a serum tube where the blood is allowed to clot. Plasma samples will be stored in ice until centrifuged twice at 1,500g for 10 minutes at 4° Celsius. Serum will be kept in room temperature for 60 minutes then centrifuged at 1300g for 10 minutes. Both samples will be divided into separate 1.8-mL microcentrifuge tubes and will be frozen at -80° C for later analysis.
Change in stroke volume | Baseline to twelve weeks
  Participants will wear an FDA approved wristwatch (Biobeat technologies, Petah Tikva, Israel) while resting in a seated position. Measurements will be taken in an urgent mode - every minute for five minutes.
Change in fat percentage | Baseline to twelve weeks
  Fat percent will be measured using the SECA mBCA 515 (Seca, Hamburg, Germany), a valid and reliable analyzer of body composition. Participants will drink 400 ml of water before the examination which will take place in the morning. Drinking will be stopped 30 minutes before the examination and participants will be instructed to urinate and remove any jewelries before the examination.
Change in body mass index (BMI) | Baseline to twelve weeks
  Participants' height will be measured using SECA stadiometer, and body weight will be measured using the SECA mBCA 515 (Seca, Hamburg, Germany), a valid and reliable analyzer of body composition. Participants will drink 400 ml of water before the examination which will take place in the morning. Drinking will be stopped 30 minutes before the examination and participants will be instructed to urinate and remove any jewelries before the examination.
Change in maximal muscle strength- One repetition maximum - leg curl and shoulder press | Baseline to twelve weeks
  Participants will perform a dynamic warmup including mobility and calisthenics exercises, followed by specific warm up sets of each of the exercises leg curl and shoulder press (performed on weight-stack machines). Then, up to five attempts will be made to complete one repetition sets with increasing load until the participant either fails to complete the full range of motion or declares she cannot attempt the next set. The load (in kg) of the final successful attempt for each exercise will be documented for analysis. Two to three minutes rest will be provided between the attempts. The order of the exercises will be maintained throughout the assessment points and between participants. The assessments will be carried out by the same experimenter at the same time of day ±2 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Israel Halperin, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Westcott WL. Resistance training is medicine: effects of strength training on health. Curr Sports Med Rep. 2012 Jul-Aug;11(4):209-16. doi: 10.1249/JSR.0b013e31825dabb8. PMID 22777332
- [Background] Bennie JA, De Cocker K, Smith JJ, Wiesner GH. The epidemiology of muscle-strengthening exercise in Europe: A 28-country comparison including 280,605 adults. PLoS One. 2020 Nov 25;15(11):e0242220. doi: 10.1371/journal.pone.0242220. eCollection 2020. PMID 33237930
- [Background] Phillips SM, Winett RA. Uncomplicated resistance training and health-related outcomes: evidence for a public health mandate. Curr Sports Med Rep. 2010 Jul-Aug;9(4):208-13. doi: 10.1249/JSR.0b013e3181e7da73. PMID 20622538
- [Background] Iwatsuki T, Abdollahipour R, Psotta R, Lewthwaite R, Wulf G. Autonomy facilitates repeated maximum force productions. Hum Mov Sci. 2017 Oct;55:264-268. doi: 10.1016/j.humov.2017.08.016. Epub 2017 Sep 1. PMID 28865313
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Helms ER, Byrnes RK, Cooke DM, Haischer MH, Carzoli JP, Johnson TK, Cross MR, Cronin JB, Storey AG, Zourdos MC. RPE vs. Percentage 1RM Loading in Periodized Programs Matched for Sets and Repetitions. Front Physiol. 2018 Mar 21;9:247. doi: 10.3389/fphys.2018.00247. eCollection 2018. PMID 29628895
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893